CLINICAL TRIAL: NCT03101592
Title: INTERVAL: Varying Intervals of ART to Improve Outcomes in HIV
Acronym: INTERVAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment completed. Outcomes measured after only 1 yr due to loss of funding.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Boston University (Other); Equip, Lesotho (Other); Ministry of Health, Malawi (Other Government); Ministry of Health, Zambia (Other Government); Partners in Hope, Inc. (Industry); Right to Care (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Risa Hoffman, MD, MPH, Associate Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-001652
Record Dates: First submitted 2017-03-18; First posted 2017-04-05 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: HIV-1-infection
Keywords: antiretroviral therapy; retention; ART; cost-effectiveness; virologic suppression

STUDY DESIGN:
Intervention Model Description: The study will be a cluster randomized trial comparing three different antiretroviral therapy (ART) dispensing strategies. Clusters will be comprised of individual clinics in Malawi and Zambia. Enrolled individuals will receive standard of care at their site with the exception of the ART dispensing interval based on the assigned randomization. Outcomes will be assessed after 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care ART dispensing (No Intervention): The standard of care arm will allow ART dispensing based on usual practice at the clinic. Standard of care is anticipated to have variability in how ART is dispensed, although the approach should be consistent with applicable country guidelines at the time of study.
- Three-month ART dispensing (Experimental): Providers at facilities randomized to three-month ART dispensing will be expected to provide all enrolled patients with a 90-day supply of ART and associated HIV medications (cotrimoxazole and isoniazid if part of country guidelines). All other aspects of care will be as per standard of care for the enrolling clinic.
  Interventions: Other: Three-month ART dispensing
- Six-month ART dispensing (Experimental): Providers at facilities randomized to six-month ART dispensing will be expected to provide all enrolled patients with a 180-day supply of ART and associated HIV medications (cotrimoxazole and isoniazid if part of country guidelines). All other aspects of care will be as per standard of care for the enrolling clinic.
  Interventions: Other: Six-month ART dispensing

INTERVENTIONS:
Other: Three-month ART dispensing — Patients enrolled in the three-month ART dispensing arm will receive a 90-day supply of ART from their provider for the duration of the study.
  Arms: Three-month ART dispensing
Other: Six-month ART dispensing — Patients enrolled in the six-month ART dispensing arm will receive a 180-day supply of ART from their provider for the duration of the study.
  Arms: Six-month ART dispensing

SUMMARY:
This is an unblinded cluster-randomized study to evaluate the effectiveness of two strategies for scripting/dispensing of antiretroviral therapy (ART) on retention, virologic suppression, and cost compared to the standard of care. The study will be conducted in Malawi and Zambia among approximately 8,200 HIV-1-infected adults (18 years or older) who are stable on ART. Clusters will be randomized to one of three study arms: (1) standard of care (SOC) ART scripting (varies by country, region, clinic, and/or provider), (2) three-month ART scripting, and (3) six-month ART scripting. 30 clusters will be selected for the study, 15 in Malawi and 15 in Zambia, and will be randomized to a study arm.

DETAILED DESCRIPTION:
This study will be conducted among approximately 8,200 HIV-infected individuals age 18 years or older who are stable on antiretroviral therapy (ART) in 30 clusters in Malawi and Zambia. Individuals will be screened at routine clinic visits and enrolled if they meet inclusion criteria. Enrolled individuals will receive standard of care at their site with the exception of their ART dispensing interval based on the assigned randomization. Outcomes will be assessed after 12 months, but all participants will be under observational follow-up for 36 months, with annual re-assessment of retention, virologic suppression, and cost-effectiveness.

There will be no contact with study participants during the period of follow-up.

Endpoints will be determined by chart review after the primary endpoint is reached (12 months). Endpoint data collection will include:

1. Retention in care on strategy
2. Suppressed viral load of <1,000 copies done as part of standard of care viral load monitoring

In a subset of participants in Malawi (n=1,500), we will perform a review of participants' health passports, a record of patient clinic visits, general health information, and medications that is possessed by patients in Malawi, after the 12-month endpoint has been completed. Data will be collected on interim clinic visits, such as reason for visit/services received (sick, family planning, non-communicable disease treatment), frequency of visits, and location of clinic services.

In a subset of participants (~240), we will perform a post intervention study visit after the 12-month endpoint is completed. Qualitative interviews will be performed with a subset of participants and will focus on patient experience with assigned dispensing interval, including challenges/barriers and facilitators towards adherence and retention. Focused questions around endpoints (if default, reasons; if virologic failure, reasons including adherence) will also be addressed in the post-intervention visit.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Willing and able to provide written informed consent for participation in this study.
* Confirmed HIV-1 infection based on country standard of care for testing.
* On antiretroviral treatment (ART) for at least six months.
* On a first-line ART regimen as defined by country-specific guidelines.
* No drug toxicity/tolerability issues with ART regimen within the prior six months.
* No period of more than one month without ART medication possession within the last six months.
* No active opportunistic infection suspected (including tuberculosis) and not treated for an opportunistic infection in the last 30 days.
* No active comorbidity (including hypertension) and not treated for a comorbidity in the last 30 days.
* No viral load of more than 1000 copies/ml (using standard assay) within the last six months.
* Not currently pregnant.
* At least six months postpartum if recently delivered a baby.
* Not currently breastfeeding or planning to breastfeed.

Exclusion Criteria:

* Under 18 years of age.
* Viral load of 1000 copies/ml or greater (using standard assay) within the last six months.
* On alternative first-line or second-line ART regimen.
* One month or more without medication possession within the last six months.
* Experienced an ART toxicity/tolerability issue within the last six months.
* Currently receiving treatment for tuberculosis or receiving treatment for any other opportunistic infection or comorbidity (including hypertension).
* Pregnant or less than six months postpartum.
* Women who are breastfeeding.
* Unwilling or unable to provide informed consent.
* Previously enrolled in the study.
* Currently enrolled in any other research study at the site that involves adherence/retention or alters delivery of HIV care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9118 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Risa M Hoffman, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (2):
- Partners in Hope, Lilongwe, Malawi
- EQUIP Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffman RM, Moyo C, Balakasi KT, Siwale Z, Hubbard J, Bardon A, Fox MP, Kakwesa G, Kalua T, Nyasa-Haambokoma M, Dovel K, Campbell PM, Tseng CH, Pisa PT, Cele R, Gupta S, Benade M, Long L, Xulu T, Sanne I, Rosen S. Multimonth dispensing of up to 6 months of antiretroviral therapy in Malawi and Zambia (INTERVAL): a cluster-randomised, non-blinded, non-inferiority trial. Lancet Glob Health. 2021 May;9(5):e628-e638. doi: 10.1016/S2214-109X(21)00039-5. PMID 33865471
- [Derived] Phiri K, McBride K, Siwale Z, Hubbard J, Bardon A, Moucheraud C, Haambokoma M, Pisa PT, Moyo C, Hoffman RM. Provider experiences with three- and six-month antiretroviral therapy dispensing for stable clients in Zambia. AIDS Care. 2021 Apr;33(4):541-547. doi: 10.1080/09540121.2020.1755010. Epub 2020 May 4. PMID 32363910
- [Derived] Hoffman R, Bardon A, Rosen S, Fox M, Kalua T, Xulu T, Taylor A, Sanne I. Varying intervals of antiretroviral medication dispensing to improve outcomes for HIV patients (The INTERVAL Study): study protocol for a randomized controlled trial. Trials. 2017 Oct 13;18(1):476. doi: 10.1186/s13063-017-2177-z. PMID 29029644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment relied on active identification and referral of stable patients by clinic staff. Clinics were randomized to a study arm, and enrolled individuals initiated the study drug dispensing interval to which the clinic had been randomly assigned.
  A total of 14,430 individuals were screened from May 2017- April 2018 across 30 study sites.
Units Other Than Participants: clinics
Period: Overall Study
Arm/Group | Standard of Care ART Dispensing | Three-month ART Dispensing | Six-month ART Dispensing
Started | 3123; 10 clinics | 2896; 10 clinics | 3099; 10 clinics
Completed | 3012; 10 clinics | 2726; 10 clinics | 2981; 10 clinics
Not Completed | 111; 0 clinics | 170; 0 clinics | 118; 0 clinics
Not completed — participant files could not be located | 111 | 170 | 118

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized for just the participants for whom endpoint data was available. 399 participant files could not be located for recording outcome data, so they were excluded from these analyses.
Units Other Than Participants: clinics
Groups:
- Standard of Care ART Dispensing (SOC): The standard of care arm will allow ART dispensing based on usual practice at the clinic. Standard of care is anticipated to have variability in how ART is dispensed, although the approach should be consistent with applicable country guidelines at the time of study.
- Three-month ART Dispensing (3MD): Providers at facilities randomized to three-month ART dispensing will be expected to provide all enrolled patients with a 90-day supply of ART and associated HIV medications (cotrimoxazole and isoniazid if part of country guidelines). All other aspects of care will be as per standard of care for the enrolling clinic.
  Three-month ART dispensing: Patients enrolled in the three-month ART dispensing arm will receive a 90-day supply of ART from their provider for the duration of the study.
- Six-month ART Dispensing (6MD): Providers at facilities randomized to six-month ART dispensing will be expected to provide all enrolled patients with a 180-day supply of ART and associated HIV medications (cotrimoxazole and isoniazid if part of country guidelines). All other aspects of care will be as per standard of care for the enrolling clinic.
  Six-month ART dispensing: Patients enrolled in the six-month ART dispensing arm will receive a 180-day supply of ART from their provider for the duration of the study.
- Total: Total of all reporting groups
Arm/Group | Standard of Care ART Dispensing (SOC) | Three-month ART Dispensing (3MD) | Six-month ART Dispensing (6MD) | Total
Number analyzed (Participants) | 3012 | 2726 | 2981 | 8719
Number analyzed (clinics) | 10 | 10 | 10 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: For each demographic variable analyzed, some responses were missing, so could not be included.
  years
    number analyzed (Participants) | 2965 | 2669 | 2956 | 8590
    (all) | 42.9 [35.9 to 50.3] | 42.7 [36.1 to 49.6] | 42.6 [36.2 to 49.7] | 42.6 [35.9 to 49.8]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In the SOC arm, there was 1 missing data point for sex.
  Participants
    number analyzed (Participants) | 3011 | 2726 | 2981 | 8718
    Female | 2020 | 1841 | 1913 | 5774
    Male | 991 | 885 | 1068 | 2944
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    (all) |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 1532 | 1430 | 1588 | 4550
  Zambia | 1480 | 1296 | 1393 | 4169
Disclosure of HIV status to primary partner [Count of Participants; unit: Participants] — Population: The number that disclosed HIV status was among those who reported having a primary partner. Additionally, there were missing/not answered data for each arm: in the standard of care arm, 3 were missing; in 3MD 3 were missing; and in 6MD, 1 was missing.
  Participants
    number analyzed (Participants) | 2215 | 2043 | 2266 | 6524
    Yes | 2054 | 1819 | 2100 | 5973
    No | 161 | 224 | 166 | 551
Median years on ART [Median (Inter-Quartile Range); unit: years] — Population: Medians calculated among those with data available
  years
    number analyzed (Participants) | 2030 | 1666 | 1885 | 5581
    (all) | 4.9 [2.6 to 8.4] | 5.4 [2.8 to 8.2] | 4.9 [2.6 to 7.9] | 5.0 [2.7 to 8.2]
Marital status [Count of Participants; unit: Participants] — Population: In the 3MD arm and 6MD arm, there was 1 missing from each.
  Participants
    number analyzed (Participants) | 3012 | 2725 | 2980 | 8717
    Married or long-term partner | 1889 | 1650 | 1977 | 5516
    Single or no long-term partner | 247 | 248 | 267 | 762
    Widowed, divorced, or separated | 876 | 827 | 736 | 2439
Median household size [Median (Inter-Quartile Range); unit: People in household] — Population: Calculated by arm and overall
  People in household | 4 [3 to 6] | 5 [3 to 6] | 5 [3 to 6] | 4 [3 to 6]
School (highest level completed) [Count of Participants; unit: Participants] — Population: Missing/not answered: SOC arm- 7; 3MD arm- 4; 6MD arm- 17
  Participants
    number analyzed (Participants) | 3005 | 2722 | 2964 | 8691
    No education or less than primary school | 574 | 480 | 347 | 1401
    Primary school | 1453 | 1293 | 1372 | 4118
    Secondary school | 841 | 811 | 978 | 2630
    University/Graduate | 137 | 138 | 267 | 542
Work status [Count of Participants; unit: Participants] — Population: 6 missing/not answered from the SOC arm, 4 from the 3MD arm, and 4 from the 6MD arm
  Participants
    number analyzed (Participants) | 3006 | 2722 | 2977 | 8705
    Formal employment | 450 | 398 | 629 | 1477
    Informal employment | 1435 | 1027 | 1545 | 4007
    Not working | 1121 | 1297 | 803 | 3221
Missed work to attend current ART clinic visit [Count of Participants; unit: Participants] — Population: Missing/Unanswered for SOC arm = 8, 3MD arm = 6, 6MD arm =4.
  Participants
    number analyzed (Participants) | 3004 | 2720 | 2977 | 8701
    (all) | 1490 | 1101 | 1600 | 4191
Average monthly earnings [Median (Inter-Quartile Range); unit: USD] — Population: Average monthly earnings among those who reported working in US dollars
  USD
    number analyzed (Participants) | 1861 | 1418 | 2158 | 5437
    (all) | 48.02 [13.80 to 138.00] | 66.24 [19.32 to 198.78] | 72.45 [27.60 to 198.78] | 60.00 [20.00 to 186.1]
Transport method to ART clinic [Count of Participants; unit: Participants]
  Walk | 1786 | 1618 | 1306 | 4710
  Bicycle | 339 | 304 | 385 | 1028
  Bus or minibus | 770 | 634 | 925 | 2329
  Bicycle taxi | 65 | 96 | 237 | 398
  Personal or friend's vehicle | 42 | 55 | 119 | 216
  Other | 10 | 19 | 9 | 38
Median one-way travel time to clinic [Median (Inter-Quartile Range); unit: minutes] — Population: Medians overall and by arm among those for whom data were reported.
  minutes | 40.2 [19.8 to 66.5] | 45.0 [25.2 to 90.0] | 40.2 [19.8 to 60.0] | 40.3 [20.0 to 80.0]
Proportion of patients incurring transport costs to clinic [Count of Participants; unit: Participants] | 917 | 812 | 1265 | 2994
For those incurring transport costs, median one-way cost [Median (Inter-Quartile Range); unit: USD] — Population: For those who did incur transport costs.
  USD
    number analyzed (Participants) | 917 | 812 | 1265 | 2994
    (all) | 0.69 [0.30 to 1.0] | 0.55 [0.40 to 0.97] | 0.69 [0.41 to 1.38] | 0.69 [0.40 to 1.11]
Median time spent at ART clinic [Median (Inter-Quartile Range); unit: minutes] — Population: Medians by arm and overall.
  minutes | 120.0 [60.0 to 180.0] | 180.0 [120.0 to 240.0] | 180.0 [120.0 to 240.0] | 150.0 [90.0 to 240.0]
Median ART dispensing interval in year prior [Median (Inter-Quartile Range); unit: days] — Population: Medians by arm and overall
  days
    number analyzed (Participants) | 2208 | 2084 | 2197 | 6489
    (all) | 60.0 [43.0 to 90.0] | 80.0 [60.0 to 90.0] | 78.0 [60.0 to 90.0] | 75.0 [54.0 to 90.0]
Among reproductive age women, received contraception in last three months [Count of Participants; unit: Participants] — Population: This variable was just among women of reproductive age. In each arm, there were missing/unanswered among this group: in the SOC arm= 204, 3MD arm = 212, 6MD arm = 220.
  Participants
    number analyzed (Participants) | 1001 | 962 | 1035 | 2998
    (all) | 139 | 155 | 214 | 508

OUTCOME MEASURES:

1. Primary Outcome: Retention in Care at 12 Months
Description: The primary outcome to be studied is whether scripting/dispensing of ART for intervals of six months is non-inferior to three months with respect to retention in care.
Time Frame: 12 months
Population: The sample includes only those participants for whom outcome data was available (n=8719). As described in the participant flow, 399 participant files could not be located to analyze final outcome data at the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care ART Dispensing (SOC) | Three-month ART Dispensing (3MD) | Six-month ART Dispensing (6MD)
Number analyzed (Participants) | 3012 | 2726 | 2981
Participants
  Retention | 2478 | 2356 | 2729
  Transfer | 60 | 66 | 58
  Death | 11 | 8 | 8
  Lost to follow-up | 463 | 296 | 186
Statistical Analysis 1: Comparison: Standard of Care ART Dispensing (SOC) vs Three-month ART Dispensing (3MD); Our sample size was estimated for a cluster-randomized non-inferiority trial. We had 30 clusters available for randomization and assumed a fixed number of clusters (k), an equal number of clusters per arm, and an equal number of subjects per cluster; Test type: Non-Inferiority — We estimated that approximately 5% of subjects would fail to be retained in care in the standard of care arm, and a retention rate <7·5% to be non-inferior in the three-month or six-month study arms, with a 2·5% non-inferiority margin. Assuming an alpha of 0.05, power of 90%, and an intracluster correlation coefficient (ICC) of 0·004, we estimated a sample size of 271 subjects per cluster for a total of 2,710 subjects per arm and 8,130 total individuals; Risk Difference (RD) = 4.0, 95% CI 2-sided [-4.3 to 12.3] — RD is for retention 3MD vs. SOC
Statistical Analysis 2: Comparison: Standard of Care ART Dispensing (SOC) vs Six-month ART Dispensing (6MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 9.1, 95% CI 2-sided [0.9 to 17.2] — RD is for retention 6MD vs. SOC
Statistical Analysis 3: Comparison: Three-month ART Dispensing (3MD) vs Six-month ART Dispensing (6MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 5, 95% CI 2-sided [1 to 9.1] — RD is for retention 6MD vs. 3MD
Statistical Analysis 4: Comparison: Standard of Care ART Dispensing (SOC) vs Three-month ART Dispensing (3MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.4, 95% CI 2-sided [-0.8 to 1.6] — RD is for transfer 3MD vs. SOC
Statistical Analysis 5: Comparison: Standard of Care ART Dispensing (SOC) vs Six-month ART Dispensing (6MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.1, 95% CI 2-sided [-0.9 to 0.8] — RD is for transfer 6MD vs. SOC
Statistical Analysis 6: Comparison: Three-month ART Dispensing (3MD) vs Six-month ART Dispensing (6MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.5, 95% CI 2-sided [-1.7 to 0.7] — RD is for transfer 6MD vs. 3MD
Statistical Analysis 7: Comparison: Standard of Care ART Dispensing (SOC) vs Three-month ART Dispensing (3MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.1, 95% CI 2-sided [-0.4 to 0.2] — RD is for death 3MD vs. SOC
Statistical Analysis 8: Comparison: Standard of Care ART Dispensing (SOC) vs Six-month ART Dispensing (6MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -0.1, 95% CI 2-sided [-0.9 to 0.8] — RD is for death 6MD vs. SOC
Statistical Analysis 9: Comparison: Three-month ART Dispensing (3MD) vs Six-month ART Dispensing (6MD); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.0, 95% CI 2-sided [-0.3 to 0.3] — RD is for death 6MD vs. 3MD

2. Secondary Outcome: Virologic Suppression at 12 Months
Description: The secondary outcome to be studied is whether scripting/dispensing of ART for intervals of six months is non-inferior to three months with respect to a viral load outcome of <1,000 copies/ml (undetectable) at 12 months.
Time Frame: 12 months
Population: Viral load was originally listed as a secondary outcome. However, given the nature of this implementation science project, and under real world conditions, Viral Load testing was not done due to the early state of viral load scale-up in both Malawi and Zambia.
Arm/Group | Standard of Care ART Dispensing (SOC) | Three-month ART Dispensing (3MD) | Six-month ART Dispensing (6MD)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Provider Cost Per Patient by Outcome (USD) (Mean, 95% CI)
Description: The secondary outcome to be studied is the cost-effectiveness of scripting/dispensing of ART for intervals of six months compared to three months and SOC. Cost-effectiveness will be estimated as the average cost per successful outcome (patient retained at 12 months).
Time Frame: 12 months
Population: For the cost analysis, we excluded 179 participants whose visit data were unclear, leaving an analytic sample of 8,540 patients.
Measure: Mean (95% Confidence Interval); unit: US Dollars
Groups:
- Malawi: Standard of Care (SOC): Patients in the standard of care arm in Malawi.
- Malawi: 3 Month Dispensing (3MD): Patients in the 3 month dispensing arm in Malawi.
- Malawi: 6 Month Dispensing (6MD): Patients in the 6 month dispensing arm in Malawi.
- Zambia: Standard of Care (SOC): Patients in the standard of care arm in Zambia.
- Zambia: 3 Month Dispensing (3MD): Patients in the 3 month dispensing arm in Zambia.
- Zambia: 6 Month Dispensing (6MD): Patients in the 6 month dispensing arm in Zambia.
Arm/Group | Malawi: Standard of Care (SOC) | Malawi: 3 Month Dispensing (3MD) | Malawi: 6 Month Dispensing (6MD) | Zambia: Standard of Care (SOC) | Zambia: 3 Month Dispensing (3MD) | Zambia: 6 Month Dispensing (6MD)
Number analyzed (Participants) | 1328 | 1224 | 1465 | 1101 | 1056 | 1241
US Dollars
  Achieved primary outcome | 89.00 [87.90 to 91.90] | 88.40 [86.44 to 90.36] | 85.92 [83.97 to 87.89] | 143.60 [141.68 to 145.60] | 141.60 [139.64 to 143.56] | 131.13 [129.20 to 133.12]
  Did not achieve primary outcome | 63.40 [61.42 to 65.37] | 62.30 [60.35 to 64.30] | 66.10 [64.12 to 68.09] | 99.00 [97.04 to 100.98] | 99.00 [97.04 to 100.98] | 99.00 [96.98 to 100.92]
  All patients | 86.50 [84.50 to 88.42] | 86.00 [83.99 to 87.91] | 84.60 [82.62 to 86.54] | 132.00 [130.43 to 134.35] | 134.00 [132.09 to 136.02] | 128.00 [125.64 to 129.57]

ADVERSE EVENTS:
Time Frame: From enrollment through 1 year of follow-up with all participants
Arm/Group | Standard of Care ART Dispensing (SOC) | Three-month ART Dispensing (3MD) | Six-month ART Dispensing (6MD)
All-Cause Mortality (participants affected / at risk) | 11/3012 | 8/2726 | 8/2981
Serious Adverse Events (participants affected / at risk) | 0/3012 | 0/2726 | 0/2981
Other Adverse Events (participants affected / at risk) | 0/3012 | 0/2726 | 0/2981

LIMITATIONS AND CAVEATS:
As an implementation science study of service delivery, we faced limitations common in real-world interventions. Most participants did not have routine viral load tests and funding limitations reduced the follow-up period to one year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03101592/Prot_SAP_000.pdf